CLINICAL TRIAL: NCT04004741
Title: Effects of Osteopathic Manipulative Therapy on Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1464
Record Dates: First submitted 2019-06-17; First posted 2019-07-02 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Arrhythmia
Keywords: Osteopathic Manipulative Medicine
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): Group A will receive osteopathic treatment by NMM/OMM board certified attending physicians. The protocol for the OMT intervention group is based on the guidelines set forth previously in textbooks. The protocol will last 25 minutes total, with 10 minutes for the evaluation and 15 minutes for treatment. The protocol will start in ribs so as to not exacerbate any tachyarrhythmias with rib raising, thoracic myofascial release, and a pectoralis lift. The investigator will then proceed with opening the thoracic inlet, cervical myofascial release, suboccipital release, and then end by checking for and treating Chapman's points. The physician will submit their osteopathic evaluation and fill out a form in order to determine if certain arrhythmias have an associated trigger point.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Light Touch Treatment (Sham Comparator): Group B will receive a light touch treatment, based on previous research done studying heart rate variability and OMM, where sham treatment was utilized. The protocol consisted of contacting the right ankle, left knee, right hip, diaphragm, right shoulder, neck, and cranium for precisely two minutes each, with the goal of preventing placebo autonomic nervous system stimulation. The protocol is 25 minutes long, with 10 minutes for the evaluation and 15 minutes for treatment.
  Interventions: Procedure: Light Touch Therapy

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — The purpose of this research is to investigate the effect of osteopathic manipulative treatment (OMT) focused on somatic dysfunctions commonly associated with arrhythmias on the amount of quantifiable arrhythmias as recorded on a diagnostic device.
  It is known that OMT has a stabilizing effect on the autonomic nervous system, which plays a key role in regulating heart rate and blood pressure. This increases parasympathetic tone and decreases sympathetic tone, which generally stabilizes the heart with an antiarrhythmic effect.
  Previous work has been done showing that osteopathic treatment is a beneficial adjunctive therapy for paroxysmal atrial fibrillation and decreased symptoms, though has not been proven to be helpful for patients with heart failure.
  While the effect of OMT on the neurology has been studied, we would like to further research the effect OMT specifically has on arrhythmias using more quantifiable data from implanted devices.
  Arms: Osteopathic Manipulative Treatment
Procedure: Light Touch Therapy — The physician will contact various areas of the body for 120 seconds each to expose the subject to a similar environment as the interventional group, without stimulating the autonomic nervous system.
  Arms: Light Touch Treatment

SUMMARY:
The study focuses on patients who have already been diagnosed with an arrhythmia. This is a randomized control trial that will use measurements from the implanted devices to quantify changes in the number of cardiac events experienced. Subjects will present to the Long Island Heart Rhythm Clinic (LIHRC) at the New York Institute of Technology (NYIT) Academic Health Care Center for their scheduled appointment with Dr. Cohen. These patients are generally coming in for their electrophysiology cardiology checkup, postsurgical visit, or consultation concerning their cardiac health. Once confirmed the patients meet the inclusion criteria, they will be informed about this proposed study and asked if they would like to participate. They will then be consented and randomized according to the randomization procedure outlined below.

Once enrolled, the patients will complete the study as outlined in the procedures below. They will have a baseline EKG taken, and then proceed to either Osteopathic manipulative medicine (OMM) treatment or control somatic dysfunction (SD) evaluation. The investigators will then analyze the CareLink data, or the web-based management service for the respective device, to quantify the effects the OMM or control SD evaluation had on any arrhythmia events.

All investigators delivering OMM will be neuromuscular medicine/osteopathic manipulative medicine (NMM/OMM) board certified attending physicians and trained in the specific techniques that have been associated with arrhythmia SDs and treatment modalities to have consistency when treating subjects. Subject confidentiality will be maintained throughout the process as delineated in Question 5 of the protocol document.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject has an implanted device connected to CareLink, Merlin, or respective web-based monitoring device, for at least one month
* Subject has documented diagnosis of a controlled arrhythmia
* If subject has been prescribed anticoagulants, the patients has been taking them for at least one month prior to intervention

Exclusion Criteria:

* Subject planning any surgeries, device updates or changes in the next month
* Subject's treatment regimen, including any medications, will be changed in next month
* Subject has contraindications to undergo OMT, which include prior spinal surgery, prior spinal fracture, any acute fractures over regions being treated or open wounds, current infection, or any other medical conditions that would prohibit OMT
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Decrease in Cardiac Events | 1 month from enrollment.
  The authors believe that OMT will change the number of cardiac events in arrhythmic patients, as measured on CareLink system for those with Medtronic devices, or the comparable online system for the other various manufacturers as detailed below, via the patient's implanted devices.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Cohen, MD, Principal Investigator — New York Institute of Technology College of Osteopathic Medicine
Locations (1):
- New York Institute of Technology's Academic Health Care Center, Glen Head, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomaz SR, Teixeira FA, de Lima ACGB, Cipriano Junior G, Formiga MF, Cahalin LP. Osteopathic manual therapy in heart failure patients: A randomized clinical trial. J Bodyw Mov Ther. 2018 Apr;22(2):293-299. doi: 10.1016/j.jbmt.2017.07.011. Epub 2017 Jul 29. PMID 29861222
- [Background] Fu DG. Cardiac Arrhythmias: Diagnosis, Symptoms, and Treatments. Cell Biochem Biophys. 2015 Nov;73(2):291-296. doi: 10.1007/s12013-015-0626-4. PMID 25737133
- [Background] Kirchhof P. The future of atrial fibrillation management: integrated care and stratified therapy. Lancet. 2017 Oct 21;390(10105):1873-1887. doi: 10.1016/S0140-6736(17)31072-3. Epub 2017 Apr 28. PMID 28460828
- [Background] Berger M, Schweitzer P. Timing of thromboembolic events after electrical cardioversion of atrial fibrillation or flutter: a retrospective analysis. Am J Cardiol. 1998 Dec 15;82(12):1545-7, A8. doi: 10.1016/s0002-9149(98)00704-8. PMID 9874066
- [Result] Ruffini N, D'Alessandro G, Mariani N, Pollastrelli A, Cardinali L, Cerritelli F. Variations of high frequency parameter of heart rate variability following osteopathic manipulative treatment in healthy subjects compared to control group and sham therapy: randomized controlled trial. Front Neurosci. 2015 Aug 4;9:272. doi: 10.3389/fnins.2015.00272. eCollection 2015. PMID 26300719
- [Derived] Nikakis J, Tale E, Malkov D, Arora US, Keys J, Li TS, Yao SC, Cohen TJ. The effect of osteopathic manipulative treatment on quality of life in patients with cardiac implantable electronic devices. J Osteopath Med. 2024 Apr 19;124(8):365-368. doi: 10.1515/jom-2023-0218. eCollection 2024 Aug 1. PMID 38632892